CLINICAL TRIAL: NCT02134912
Title: S1300: A Randomized, Phase II Trial of Crizotinib Plus Pemetrexed Versus Pemetrexed Monotherapy in ALK-Positive Non-squamous NSCLC Patients Who Have Progressed Systemically After Previous Clinical Benefit From Crizotinib Monotherapy
Brief Title: S1300: Pemetrexed Disodium With or Without Crizotinib in Treating Patients With Stage IV Non-Small Cell Lung Cancer That Has Progressed After Crizotinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: science has moved forward and there is no intent to complete the study
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S1300; NCI-2014-00685 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1300 (Other: SWOG); S1300 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Adenocarcinoma of the Lung; Large Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (crizotinib, pemetrexed disodium) (Experimental): Patients receive crizotinib PO BID on days 1-21 and pemetrexed disodium IV over 10 minutes on day 1.
  Interventions: Drug: crizotinib; Drug: pemetrexed disodium; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm II (pemetrexed disodium) (Experimental): ARM II: Patients receive pemetrexed disodium IV over 10 minutes on day 1. Upon disease progression or symptomatic deterioration, patients may crossover to Arm I.
  Interventions: Drug: pemetrexed disodium; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: crizotinib — Given PO
  Other Names: c-met/hepatocyte growth factor receptor tyrosine kinase inhibitor PF-02341066; c-met/HGFR tyrosine kinase inhibitor PF-02341066; MET Tyrosine Kinase Inhibitor PF-02341066; PF-02341066
  Arms: Arm I (crizotinib, pemetrexed disodium)
Drug: pemetrexed disodium — Given IV
  Other Names: ALIMTA; LY231514; MTA
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This randomized phase II trial studies how well pemetrexed disodium with or without crizotinib works in treating patients with stage IV non-small cell lung cancer that has progressed after crizotinib. Drugs used in chemotherapy, such as pemetrexed disodium, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Crizotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving pemetrexed disodium is more effective with or without crizotinib in treating patients with non-small cell lung cancer that has progressed after crizotinib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of the combination of crizotinib and pemetrexed (pemetrexed disodium) compared to pemetrexed monotherapy as measured by progression-free survival (PFS) in anaplastic lymphoma kinase (ALK)+ non-squamous non-small cell lung cancer (NSCLC) patients who achieved clinical benefit with crizotinib monotherapy and subsequently progressed systemically.

SECONDARY OBJECTIVES:

I. To compare the response rate (confirmed and unconfirmed, complete and partial responses) in patients randomized to receive pemetrexed monotherapy to historical data.

II. To assess overall survival in both arms. III. To evaluate the patterns of failure (central nervous system [CNS], extra-CNS) of the combination of crizotinib and pemetrexed and of pemetrexed monotherapy in ALK+ non-squamous NSCLC after progression on crizotinib.

IV. To evaluate the frequency and severity of toxicities resulting from the administration of crizotinib and pemetrexed compared to pemetrexed monotherapy.

V. To evaluate PFS and the response rate in patients treated with crizotinib following progression on the pemetrexed monotherapy arm.

TERTIARY OBJECTIVES:

I. To compare progression-free survival (PFS) and response rates (RR) between ALK dominant and ALK non-dominant patients in the entire study population and within each treatment arm.

II. To evaluate if the magnitude of difference in these outcomes between ALK dominant and ALK non-dominant patients varies by treatment arm.

III. To assess blood biomarkers of sensitivity and resistance to crizotinib and pemetrexed in an exploratory manner. The blood biomarkers include cell free circulating deoxyribonucleic acid (DNA), micro ribonucleic acid (microRNA) before treatment, during treatment (after 2 cycles) and at treatment progression.

IV. To assess pharmacogenomic factors in peripheral blood that might affect the drug level and treatment outcomes in an exploratory manner.

V. To assess proteomic/immunologic parameters that might affect the treatment outcomes in an exploratory manner.

VI. To evaluate the frequency of individual mechanisms of resistance (copy number gain [CNG], mutation, alternate oncogene).

VII. To identify alternative driver mechanisms in ALK fluorescence in situ hybridization positive (FISH+) otherwise unknown.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive crizotinib orally (PO) twice daily (BID) on days 1-21 and pemetrexed disodium intravenously (IV) over 10 minutes on day 1.

ARM II: Patients receive pemetrexed disodium IV over 10 minutes on day 1. Upon disease progression or symptomatic deterioration, patients may crossover to Arm I.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven primary non-squamous non-small cell lung cancer (adenocarcinoma, large cell carcinoma, adenocarcinoma in situ, mixed histology with < 50% squamous or unspecified); patients with tumors having squamous cell components >= 50% are not eligible; disease must be stage IV
* Patients must have documented ALK positivity at the time of initial crizotinib monotherapy using the Vysis Break-Apart FISH assay (or other Food and Drug Administration [FDA]-approved diagnostic test); samples are deemed to be FISH-positive if greater than or equal to 15% of scored tumor cells had split ALK 5' and 3' probe signals or had isolated 3' signal; FISH status must be documented on the Onstudy Form and a copy of the pathology report from the Vysis Break-Apart FISH assay (or other FDA-approved diagnostic test) must be submitted
* Prior to registration, patients must have achieved clinical benefit with crizotinib monotherapy and subsequently have systemically progressed; clinical benefit is defined as having stable disease on crizotinib monotherapy for at least 90 days or achieving a confirmed partial or complete response; systemic progression is defined as progressive disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, excluding progression based on brain/CNS metastases alone
* Patients must have received crizotinib monotherapy at 250 mg BID on a continuous dosing schedule for at least 90 days; patients must be planning to start treatment at least three days, but no more than 30 days after discontinuing crizotinib monotherapy; patients who were not able to tolerate 250 mg BID of crizotinib are not eligible for this study
* Patients must be pemetrexed-naïve; patients may have received any number of prior chemotherapy or molecularly targeted agents; if crizotinib was used in the 1st line setting then chemotherapy naive patients are also eligible; if patient received crizotinib in combination with chemotherapy, prior chemotherapy must have been discontinued at least 14 days prior to registration and all adverse events must have resolved to =< grade 1
* Patients must have measurable disease per RECIST documented by computed tomography (CT) or magnetic resonance imaging (MRI); the CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality; measurable disease must be assessed within 28 days prior to registration; pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease; non-measurable disease must be assessed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form RECIST 1.1
* Patients must have a CT or MRI scan of the brain to evaluate for CNS disease within 42 days prior to registration; patient must not have brain metastases unless: (1) metastases have been treated and have remained controlled for at least 14 days following treatment or was not treated, but is asymptomatic, AND (2) patient has no residual neurological dysfunction off corticosteroids or anti-convulsants for at least 14 days
* Patients may have received palliative radiotherapy to non-target lesions within 14 days prior to registration provided all radiotherapy related toxicities have resolved to =< grade 1 prior to registration; patients must not have received any major surgery within 28 days prior to registration
* Patients must not have had any prior exposure to heat shock protein (HSP)90 inhibitors (such as IPI-504 or ganetespib) or non-crizotinib ALK inhibitors (such as AP26113 or LDK378)
* Patients must be offered participation in the translational medicine studies; additionally if patient has biopsy accessible disease they must be offered participation in the translational medicine studies
* Absolute neutrophil count (ANC) >= 1,500/ul
* Platelet count >= 100,000/ul
* Hemoglobin >= 9 g/dL
* Serum bilirubin =< 2 X institutional upper limit of normal (IULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x IULN
* Estimated (calculated) or measured glomerular filtration rate >= 45 mL/min (or 45 mL/min/1.73 m^2); creatinine (mg/dl) used in calculation (Cockroft-Gault) must be obtained within 28 days prior to registration
* Male patients must have free and total testosterone level obtained within 28 days prior to registration
* Pre-study history and physical must be obtained with 28 days prior to registration
* Patients must have Zubrod performance status 0-2 within 28 days prior to registration
* Patients must be able to swallow capsules
* Patients must have corrected QT (QTC) interval =< 480 msec on electrocardiogram (EKG) at baseline; patient with congenital long QT syndrome are not eligible
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* REGULATORY CRITERIA: Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* REGULATORY CRITERIA: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* CROSSOVER (STEP 2) REGISTRATION: Patients must have progressed systemically on Arm 2 of this study (pemetrexed monotherapy)
* CROSSOVER (STEP 2) REGISTRATION: Patients must be registered to crossover (Step 2) within 30 days of discontinuing treatment on Arm 2 of this study
* CROSSOVER (STEP 2) REGISTRATION: ANC >= 1,500/ul
* CROSSOVER (STEP 2) REGISTRATION: Platelet count >= 100,000/ul
* CROSSOVER (STEP 2) REGISTRATION: Serum bilirubin =< 2 X IULN
* CROSSOVER (STEP 2) REGISTRATION: SGOT (AST) or SGPT (ALT) =< 2.5 x IULN
* CROSSOVER (STEP 2) REGISTRATION: estimated (calculated) or measured glomerular filtration rate >= 45 mL/min (or 45 mL/min/1.73 m^2) within 28 days prior to registration; creatinine (mg/dl) used in calculation (Cockroft-Gault) must be obtained within 28 days prior to registration
* CROSSOVER (STEP 2) REGISTRATION: male patients must have free and total testosterone level obtained within 28 days prior to Crossover (Step 2) Registration
* CROSSOVER (STEP 2) REGISTRATION: patients must have Zubrod performance status 0-2 within 28 days prior to Crossover (Step 2) Registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Camidge, Principal Investigator — SWOG Cancer Research Network
Locations (167):
- United States (167):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer, Sandpoint, Idaho
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Reid Health, Richmond, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Faith Regional Medical Offices West, Norfolk, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hemotology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Oncology Hematology West, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center, Scottsbluff, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Orange Regional Medical Center, Middletown, New York
  - Asheville Hematology-Oncology Associates, Asheville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - SWOG, Portland, Oregon
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There is only one patient enrolled in this study. Patient was taken off study treatment by treating physician due to recent changes in standard of care. And patient never started protocol treatment. Thus we didn't enter any results for this only patient in the trial.
Period: Overall Study
Arm/Group | Arm I (Crizotinib, Pemetrexed Disodium) | Arm II (Pemetrexed Disodium)
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The one patient that enrolled immediately withdrew consent [enrolled the day before the study closed]. No manuscript will be forthcoming.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Crizotinib, Pemetrexed Disodium) | Arm II (Pemetrexed Disodium) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: PFS Between Patients Randomized to Receive Pemetrexed Disodium Monotherapy Versus Crizotinib and Pemetrexed Disodium Combination Therapy
Description: A stratified log-rank test at the 0.10 level will be used to test the primary hypothesis comparing the two treatment arms.
Time Frame: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years
Population: as for baseline characteristics
Arm/Group | Arm I (Crizotinib, Pemetrexed Disodium) | Arm II (Pemetrexed Disodium)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Adverse Events of Crizotinib in Combination With Pemetrexed Disodium, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Comparisons of toxicities rates will be done using a Fisher's exact or chi-squared test of independence, when appropriate using 10% as the significance threshold. Within each treatment arm, any toxicity with at least 5% prevalence has at least a 95% chance of being observed.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Arm/Group | Arm I (Crizotinib, Pemetrexed Disodium) | Arm II (Pemetrexed Disodium)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Response Rate (Confirmed and Unconfirmed) With Pemetrexed Disodium Monotherapy
Description: Comparisons of response rates will be done using a chi-square test of independence using 10% as the significance threshold. Within each treatment arm, response rates can be estimated to within 13% (with 95% confidence).
Time Frame: Up to 3 years
Population: as for baseline characteristics
Arm/Group | Arm I (Crizotinib, Pemetrexed Disodium) | Arm II (Pemetrexed Disodium)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Response Rates (Confirmed and Unconfirmed) of Crizotinib With Pemetrexed Disodium
Description: as for outcome 3
Time Frame: Up to 3 years
Population: as for baseline characteristics
Arm/Group | Arm I (Crizotinib, Pemetrexed Disodium) | Arm II (Pemetrexed Disodium)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Patterns of Failure
Description: Defined as CNS-only, extra-CNS, and both CNS and extra-CNS progression between the treatment arms. Evaluated within each treatment arm using cumulative incidence curves.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Arm/Group | Arm I (Crizotinib, Pemetrexed Disodium) | Arm II (Pemetrexed Disodium)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Survival
Description: Differences in OS by treatment arm will be evaluated using a 1-sided log-rank test with significant level of 10%.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Arm/Group | Arm I (Crizotinib, Pemetrexed Disodium) | Arm II (Pemetrexed Disodium)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: The one patient that enrolled immediately withdrew consent [enrolled the day before the study closed]. No manuscript will be forthcoming.
Arm/Group | Arm I (Crizotinib, Pemetrexed Disodium) | Arm II (Pemetrexed Disodium)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The one patient that enrolled immediately withdrew consent [enrolled the day before the study closed]. No manuscript will be forthcoming.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less